CLINICAL TRIAL: NCT01341795
Title: Effect of Genetic Variation in the Transporters on Glycemic Response and Pharmacokinetics of Sitagliptin and Metformin
Brief Title: Genetic Variation in the Transporters and Hypoglycemic Agents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Doo-Yeoun Cho, Assitant Professor, Ajou University School of Medicine
Other Study IDs: GDM01
Record Dates: First submitted 2011-04-21; First posted 2011-04-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes
Keywords: Newly diagnosed type 2 diabetes patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Type 2 diabetes have become a major global health problem. Currently, metformin is used as first-line therapy in combination with lifestyle changes, and sitagliptin can be added to metformin in case of insufficient glycemic control by metformin alone, and fixed-dose combination of sitagliptin and metformin is available.

In clinical practice, inter-individual variations in response to sitagliptin and metformin treatment are commonly found, which may reflect inter-patient differences in disposition of these medications.

Sitagliptin and metformin are known as substrates of some transporters (P-gp, OAT3, OCT1 and OCT2) and some functional variations of these transporters were reported. This study is designed to clarify the effect of these transporter variants on response to sitagliptin and metformin in type 2 DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly Diagnosed Type 2 Diabetes Patients
* 20-80 years old
* Taking sitagliptin and metformin for more than 3 months

Exclusion Criteria:

* Taking other oral hypoglycemic agents
* Taking medications can induce or inhibit transporters

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly Diagnosed Type 2 Diabetes Patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-07

PRIMARY OUTCOMES:
differences of sitagliptin and metformin trough concentration according to genetic variations of transporters | After 3 months of sitagliptin and metformin treatment

SECONDARY OUTCOMES:
differences of HbA1c change according to genetic variations of transporters | Baseline and after 3 months of sitagliptin and metformin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Yeoun Cho, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea